CLINICAL TRIAL: NCT06652503
Title: The Student Wellness and Emotional Growth Resiliency (SWAG-R) Program: A 6-week Coaching Program Designed For NSU Undergraduate Students to Decrease Anxiety, Depression, and Stress and Improve Mental Health, Quality of Life, and Resiliency
Brief Title: The Student Wellness and Emotional Growth Resiliency (SWAG-R) Program
Acronym: SWAG-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-197-NSU
Record Dates: First submitted 2024-10-14; First posted 2024-10-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Depression; Stress; Wellbeing; Quality of Life
Keywords: anxiety; depression; stress; wellbeing; quality of life
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The coaching program will consist of (6) free, 60 minute online coaching sessions. You will be assigned the same coach for the 6 weeks. You can coordinate schedule day/time preferences as the sessions will be done through HIPAA Zoom. Everyone in the study will get the same coaching topics in the same order.
  Interventions: Behavioral: online mental health coaching
- Waitlist Group (No Intervention): Waitlist, no intervention group

INTERVENTIONS:
Behavioral: online mental health coaching — SWAG-R Program: A 6-week Coaching Program Designed for NSU Undergraduate Students to Decrease Anxiety, Depression, and Stress and Improve Mental Health, Quality of Life, and Resiliency
  Other Names: SWAG-R Coaching Program
  Arms: Intervention Group

SUMMARY:
The purpose of this research study is to provide a free 6-week, online psychological coaching program to NSU undergraduate students to help with anxiety, depression, and stress, while improving quality of life and healthy coping skills.

DETAILED DESCRIPTION:
* All study participants will first complete a study pre-screen over the phone with a study team member. This screening will take 10-15 minutes.
* If participants are eligible to participate in the study, participants will be verbally guided through the Informed Consent form to determine if participants have any questions. This phone call will take approximately 10 minutes.
* Participants will then be electronically sent the Informed Consent form for participant review and to complete and sign, if participants would like to participate in the study.
* Once investigators receive the signed Informed Consent document, participants will be assigned a unique Study Identification Number and first assessment measures will be sent to complete (Time Point 1). This assessment will be completed electronically at participant convenience.
* Participants will then be randomly assigned to either start the free 6-week online coaching program OR will be randomly assigned to the waitlist for 6 weeks. Participants have an equal chance of being offered the coaching program right away or being put on the waitlist.
* The coaching program will consist of (6) free, 60 minute online coaching sessions. Participants will be assigned the same coach for the 6 weeks. Participants can coordinate schedule day/time preferences as the sessions will be done through HIPAA Zoom. Everyone in the study will get the same coaching topics in the same order.
* 6 weeks later, participants will complete another assessment (Time Point 2). This assessment will be completed electronically at participant convenience.
* If participants were on the waitlist, these participants can now start the free 6 week online coaching program, if participants would like. Participants are not obligated to participate but will be offered the program.
* If participants already completed the 6 week online coaching program, participants will not have any other coaching sessions during this time.
* 6 weeks later, participants will complete another assessment (Time Point 3). This assessment will be completed electronically at participant convenience.
* 6 weeks later, participants will complete another assessment (Time Point 4). This assessment will be completed electronically at participant convenience.

ELIGIBILITY:
Inclusion Criteria:

* Currently matriculating NSU undergraduate students (ages 18+)

Exclusion Criteria:

* Students who are not current NSU undergrads, participants aged 17 and younger, students who are currently enrolled in psychotherapy or mental health services, or students with acute mental health needs (e.g., psychosis, active alcohol or substance use problems, suicidality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Participant anxiety symptom severity | From enrollment up to 24 weeks
  GAD-7 (Generalized Anxiety Disorder 7 scale): GAD-7 total score for the seven items ranges from 0 to 21.
  0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Participant depression symptoms severity | From enrollment up to 24 weeks
  PHQ-9 (Patient Health Questionnaire 9): Interpretation of Total Score 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression
Participant difficulties with emotion regulation | From enrollment up to 24 weeks
  Difficulties in Emotion Regulation Scale (DERS): a 36-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate greater difficulties in emotion regulation (i.e., greater emotion dysregulation).
Participant Stress levels | From enrollment up to 24 weeks
  Perceived Stress Scale: Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Participant Resiliency | From enrollment up to 24 weeks
  Brief Resiliency Scale: Scoring: Add the responses varying from 1-5 for all six items giving a range from 6-30. Divide the total sum by the total number of questions answered. Higher scores indicate greater resiliency.
Participant quality of life and life satisfaction | From enrollment up to 24 weeks
  WHOQOL-BREF (World Health Organization Quality of Life Brief Inventory): contains 26 items and addresses 4 QOL domains: physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items). Two other items measure overall QOL and general health.
  Items are rated on a 5-point Likert scale (low score of 1 to high score of 5) to determine a raw item score. Subsequently, the mean score for each domain is calculated, resulting in a mean score per domain that is between 4 and 20. Finally, this mean domain score is then multiplied by 4 in order to transform the domain score into a scaled score, with a higher score indicating a higher QOL.
Participant adaptive coping | From enrollment up to 24 weeks
  Brief Cope Inventory: Scales are computed as follows (with no reversals of coding):
  Self-distraction, items 1 and 19 Active coping, items 2 and 7 Denial, items 3 and 8 Substance use, items 4 and 11 Use of emotional support, items 5 and 15 Use of instrumental support, items 10 and 23 Behavioral disengagement, items 6 and 16 Venting, items 9 and 21 Positive reframing, items 12 and 17 Planning, items 14 and 25 Humor, items 18 and 28 Acceptance, items 20 and 24 Religion, items 22 and 27 Self-blame, items 13 and 26 Minimum scores on sub scales =2, maximum scores = 8 with higher scores indicating greater reliance on that type of coping.

CONTACTS AND LOCATIONS:
Overall Officials: Kayla Thayer, Ph.D., ABPP, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IDP in aggregate with the exception of any identifying participant data (i.e., participant names).